CLINICAL TRIAL: NCT00206375
Title: Concomitant Use of Growth Hormone and GnRH Agonist in Adolescent Patients With Acquired Hypothyroidism
Brief Title: Growth Hormone and GnRH Agonist in Adolescents With Acquired Hypothyroidism
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry); TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Principal Investigator, Maria Jose Redondo, Unrelated to the study: Designated by institution to enter results (Study PI is not available), Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-13213
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Growth hormone
MeSH Terms: conditions — Hypothyroidism | interventions — Growth Hormone; Human Growth Hormone; Puberty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): Group 1 will be treated only with Synthroid.
- 2 (Experimental): Group 2 will be treated with Growth hormone, synthroid, and lupron.
  Interventions: Drug: Growth hormone; Drug: Growth hormone treatment and puberty
- 3 (No Intervention): Group 3 will have acute hypothyroidism and will serve as controls.

INTERVENTIONS:
Drug: Growth hormone — Growth hormone + Synthroid + Lupron
  Other Names: Humatrope
  Arms: 2
Drug: Growth hormone treatment and puberty — Lupron once a month and growth hormone daily
  Other Names: Humatrope
  Arms: 2

SUMMARY:
The purpose of this study is to see if giving growth hormone and Lupron along with thyroid hormone will improve final height in patients with long term hypothyroidism. Lupron is a medicine which is used to delay puberty and to prevent early closure of growing bones which might increase growth potential. Growth hormone is used to restore growth rate. This study will include children with "short term" and "long term" hypothyroidism.

DETAILED DESCRIPTION:
Hypothyroidism is often associated with growth failure. It takes several years for slow growth to be noticed. This growth retardation is typically severe and progressive.

Thyroid hormone is necessary for normal growth. Treatment with thyroxine (thyroid hormone) results in rapid catch-up growth, which mostly happens during the first 18 months. Growth is accompanied by increased bone age, which means early fusion (closure of the growing bones) of the bones and reduced growth potential. For example, a patient, who is 10 years old but has bone age of 12 years, has growth potential of a 12 year old and will stop growing 2 years earlier than a 10 year old patient. According to the literature, prolonged juvenile hypothyroidism (low thyroid condition) resulted in a permanent loss in height and only 70% catch-up growth was generally achieved with thyroxine replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should have clinical and biochemical evidence of hypothyroidism, T4 less than 5.0 ng /dl , fT4 less than 1.0 mcg/dl and TSH of more than 10. Patients with prolonged hypothyroidism should have growth failure and delayed bone age of at least 2 SD from the mean. Patients with short term hypothyroidism should have normal growth velocity and bone age.
2. Females 8 to 16 years old.
3. Males 9 to 17 years old.
4. Patients without any chronic medical conditions.
5. Availability of a parent or guardian to attend study visits with the patient and to be actively involved in the patient treatment plan.
6. Give written informed consent prior to any study specific screening procedure with the understanding that the patient has the right to withdraw from the study at any time without penalty.

Exclusion Criteria:

1. Taking medications that affect their growth. (eg. Systemic corticosteroids, anabolic steroids)
2. Experiencing other health problems/conditions that affect their growth rate such as growth hormone deficiency, Cushing Syndrome, rickets, and chronic diseases.
3. Patients with any condition that is a contraindication for GH therapy would include conditions such as an active tumor, impaired glucose tolerance, neurofibromatosis (worsening of neurofibromatosis), and hypertrophy of tonsils and adenoids with sleep apnea. Contraindications for patients for GNRHa therapy would include a severe systemic reaction to GNRHa which is rare, osteopenia, and osteoporosis, because delaying puberty will worsen the condition.
4. Moving to a location that the patient will not be able to be followed by a pediatric endocrinologist.
5. Patient is not willing to continue with the study. -

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2003-05; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parvin Yazdani, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor college of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Long Term Hypothyroidism, Treated With Thyroxine Alone (Contro: Group 1 will be treated only with Synthroid. Long term hypothyroidism, treated with thyroxine alone (control group)
- Long Term Hypothyroidism, Treated With Thyroxine, GH and GnRHa: Group 2 will be treated with Growth hormone, synthroid, and lupron.
  Growth hormone: Growth hormone + Synthroid + Lupron
  Growth hormone treatment and puberty: Lupron once a month and growth hormone daily.
  Long term hypothyroidism, treated with thyroxine, GH and GnRHa
- Short Term Hypothyroidism, Treated With Thyroxine (Control 2): Group 3 will have acute hypothyroidism and will serve as controls. Short term hypothyroidism, treated with thyroxine (control group)
Period: Overall Study
Arm/Group | Long Term Hypothyroidism, Treated With Thyroxine Alone (Contro | Long Term Hypothyroidism, Treated With Thyroxine, GH and GnRHa | Short Term Hypothyroidism, Treated With Thyroxine (Control 2)
Started | 6 | 3 | 7
Completed | 3 | 1 | 3
Not Completed | 3 | 2 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3
Not completed — Study terminated due to lack of funds | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Long Term Hypothyroidism, Treated With Thyroxine Alone (Contro | Long Term Hypothyroidism, Treated With Thyroxine, GH and GnRHa | Short Term Hypothyroidism, Treated With Thyroxine (Control 2) | Total
Number analyzed (Participants) | 6 | 3 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 3 | 7 | 16
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 7 | 15
  Male | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 2 | 2 | 6 | 10
  Hispanic | 3 | 1 | 1 | 5
  Black | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0
Height (cm) [Mean (Standard Deviation); unit: cm] | 124.5 (7.2) | 121.3 (10.5) | 142.3 (11.4) | 131.7 (13.4)

OUTCOME MEASURES:

1. Primary Outcome: Final Height
Description: The study was terminated due to insufficient funds. The study was terminated and the study PI has left the institution. All efforts to locate the study PI have been exhausted and the data is no longer available and cannot be reported.
Time Frame: When bones are fused
Population: n/a. The study was terminated due to insufficient funds.The study was terminated and the study PI has left the institution. All efforts to locate the study PI have been exhausted and the data is no longer available and cannot be reported
Arm/Group | Long Term Hypothyroidism, Treated With Thyroxine Alone (Contro | Long Term Hypothyroidism, Treated With Thyroxine, GH and GnRHa | Short Term Hypothyroidism, Treated With Thyroxine (Control 2)
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Bone Age
Description: as for outcome 1
Time Frame: When bones are fused
Population: study was terminated due to insufficient funds. The study was terminated and the study PI has left the institution. All efforts to locate the study PI have been exhausted and the data is no longer available and cannot be reported
Arm/Group | Long Term Hypothyroidism, Treated With Thyroxine Alone (Contro | Long Term Hypothyroidism, Treated With Thyroxine, GH and GnRHa | Short Term Hypothyroidism, Treated With Thyroxine (Control 2)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Growth Factors
Description: as for outcome 1
Time Frame: no time frame
Population: as for outcome 2
Arm/Group | Long Term Hypothyroidism, Treated With Thyroxine Alone (Contro | Long Term Hypothyroidism, Treated With Thyroxine, GH and GnRHa | Short Term Hypothyroidism, Treated With Thyroxine (Control 2)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Long Term Hypothyroidism, Treated With Thyroxine Alone (Contro | Long Term Hypothyroidism, Treated With Thyroxine, GH and GnRHa | Short Term Hypothyroidism, Treated With Thyroxine (Control 2)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No